CLINICAL TRIAL: NCT07294079
Title: Neurocognitive Responses to Social Threat: Links to Day-to-day Connectedness and Suicidality in Adolescent Girls
Brief Title: Social Threat, Adolescent Relationships, and Suicidality Study
Acronym: STARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kiera James, Research Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25050182; K23MH141548 (NIH)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Suicidal Thoughts and Behaviors; Social Connectedness; Responses to Social Threat
Keywords: Suicide Ideation; Social Threat; EEG; Adolescent; Teen
MeSH Terms: conditions — Suicidal Ideation; Behavior

STUDY DESIGN:
Intervention Model Description: All participants will be similar (12-17 with a past year suicidal thoughts and behaviors and/or non-suicidal self-injury) and will experience the same procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents (12-17) with past year STBs and/or NSSI. (Experimental): Adolescent aged 12-17 with a past year suicidal thoughts and behaviors (STBs) and/or non-suicidal self-injury will complete an EEG task that measures their response to social threat.
  Interventions: Behavioral: Social threat

INTERVENTIONS:
Behavioral: Social threat — EEG Visit:
  Participants will be presented with pictures of female actors with emotional expressions. They will be asked to remember the identities of actors displaying happy, sad, angry, and neutral expressions and tested on their memory. This task examines participants' internal attention to facial cues of emotion while asking them to remember the identities of actors displaying emotional expressions.
  EMA Over 30 days, participants will be asked to be report on their social experiences and suicidal thoughts and behaviors three times a day.

SUMMARY:
In recent years, adolescents are having higher rates of emotional health problems, such as suicidal thoughts and behaviors (STBs). The goal of this study is to learn about how teens' attention to different types of information relates to their real-world relationships and their emotional health. The investigators hope this study will help understand why some teens go on to have suicidal thoughts and behaviors and other teens do not. This information will help investigators learn how to improve emotional health in teens and reduce teen suicides.

Participants will be 100 female adolescents (ages 12-17) at high risk for STBs who will complete a series of assessments over the course of 6 months. Assessments include a baseline clinical interview, a visit to examine neural responses during a computer tasks, daily smartphone surveys about social experiences and social connectedness, and follow up questionnaires assessing STBs. Participants will also be asked to donate their text messages during the month that they complete smartphone surveys.

The research procedures will help investigators learn how adolescents react to different types of social situations. Investigators want to see if these reactions affect:

1. How connected adolescents feel to others in their daily lives
2. Adolescents' longer-term risk for suicidal thoughts and behaviors (STBs)

Participants will be asked to:

* Complete a 10-15 minute screening call to determine eligibility for the study
* Complete one 3 hour virtual (or in-person) interview consisting of a clinical assessment and questionnaires.
* Complete a 2.5-hour in person visit to complete computer tasks while record brain signals are recorded
* Complete ~5 minute smartphone surveys three times a day for 30 days, asking about their daily social experiences and their mood and feelings.
* Provide investigators with retrospective access to their text/direct messages from the month the participant was completing the smartphone surveys.
* Complete online follow-up questionnaires at 3 and 6 months

DETAILED DESCRIPTION:
There is no assignment to conditions. All participants will receive the same intervention, which is the completion of an experimental task in which participants are asked to remember the identities of actors displaying happy, sad, angry, and neutral expressions and tested on their memory. The study is designed to evaluate the effect of sustained neurocognitive responsivity to social threat on the participants' social connectedness and suicidality.

This study includes 1) a baseline clinical interview, 2) a laboratory-based EEG assessment (which includes the experimental task described above), 3) smartphone surveys in conjunction with passive ambulatory assessment, and 4) 3- and 6-month follow-up assessments of STBs.

Specifically, after phone screening, female adolescents (n=100, ages 12-17) will complete diagnostic interviews and symptom measures to confirm eligibility. Adolescents' current and lifetime STBs, including the presence, frequency, severity, and age-of-onset of suicidal ideation, plans, behaviors, and attempts will be assessed and differentiated from non-suicidal self-injurious thoughts and behaviors using the Self-Injurious Thoughts and Behaviors Interview.

Eligible participants will be invited for a laboratory visit during which they will complete the ERP Decoding Working Memory task while EEG is recorded. During each trial of the task, a face (angry, sad, happy, neutral) is randomly presented in the center of the screen. Participants are asked to remember the identity of the actor and will be tested on their memory of the identity after a delay. Specifically, participants will be asked to identify the actor from a group of four actors displaying the same emotion.

Following the laboratory visit, adolescents will complete 30-days of smartphone surveys (i.e., ecological momentary assessments [EMA]; 3 samples/day) assessing social experiences, social connectedness, and STBs. Following standard procedures, they will be randomly sampled within three blocks of time (morning, after school, evening) for a total of 90 surveys. Youth can "snooze" each prompt for up to one hour. The after-school prompt allows youth to report on experiences and thoughts they had during the school day. Once a week during the 30-day EMA protocol, participants will complete questions assessing STBs currently and during the previous week, using items adapted for EMA from the Columbia-Suicide Severity Rating Scale. During these weekly assessments, participants will indicate any STBs in the last week (i.e., since the last assessment). Finally, participants' time-stamped text, iMessage, and WhatsApp messaging logs will be downloaded at the end of the 30-day period using the software, iMazing, which creates an encrypted backup of these data.

Finally, STB assessments will be repeated at the 3- and 6-month follow-up assessments.

Certain information is withheld to protect the scientific integrity of the study design.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 12-17
* Reported recurrent suicidal thoughts and behaviors and/or non-suicidal self-injury within the past year.
* Medically and neurologically healthy, including no evidence of intellectual disability or serious cognitive impairment that would interfere with task performance
* Assigned female at birth
* Willing and able to give informed assent
* Own an iPhone

Exclusion Criteria:

* Unable to read or speak English or cognitive impairment preventing ability to complete assessments
* Lifetime presence of a neurological or serious medical condition
* Lifetime presence of a DSM-5 Autistic Spectrum Disorder
* Current DSM-5 Psychotic Disorder or severe Substance Use Disorder
* Uncorrected visual disturbance (<20/40 Snellen visual acuity)
* Presence of head injury or congenital neurological anomalies (based on parent report).

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Day-to-day social connectedness | 1 month
  Participants will be asked to rate their social connectedness with their parents/caregivers and peers 3x a day for 30 days using a 0 (not connected) to 100 (very connected) point scale.
Suicidal thoughts and behaviors | 1, 2, 3, and 4 weeks after the intervention as well as three and six months later
  Participants' suicidal thoughts and behaviors will be assessed will be assessed using the Self-Injurious Thoughts and Behaviors Interview (SITBI) and Suicidal Ideation Questionnaire-Jr (SIQ-JR). Severity of suicidal thoughts and behaviors will be operationalized as (0) absent, (1) passive SI, (2) active SI, (3) SI with a method, (4) SI with some intent, but no specific plan, (5) SI with specific plan and intent, and (6) suicide attempt(s).

CONTACTS AND LOCATIONS:
Overall Officials: Kiera M James, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the study, after deidentification, may be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Scientific data will be made accessible no later than 1 year after the grant end date. Any subject level data and associated analyzed data will be shared at time of publication. No end date.
Access Criteria: Deidentified data will be submitted to and made available on the National Institute of Mental Health Data Archive (NDA). To obtain data access, researchers will follow the established procedures within NDA, and the NDA Data Access Committee will determine the approvals for these requests. Access will be given for any legitimate scientific purpose, as determined by NDA Access Committee.